CLINICAL TRIAL: NCT06797570
Title: Nocebo Effecten Verminderen in Kinderen Met ADHD: the NOVA Study
Brief Title: The Primary Objective of This Study is to Determine Whether Positively Framed Information (PFI) on Side Effects, Compared to Negatively Framed and Extensive Information (NFI) Can Reduce the Number and Severity of Reported Adverse Events Caused by ADHD Medication in Children Aged 7 to 17 Years.
Acronym: NOVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Dunya Seinen, Student investigator medicine, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R&D/Z24.090
Record Dates: First submitted 2025-01-16; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Attention Deficit Disorder; Attention Deficit Disorder (ADD); Attention Deficit Disorder with Hyperactivity; ADHD; ADD; ADHD-not Other Specified; ADHD or ADHD Traits; ADHD Predominantly Hyperactivity Type; ADHD Predominantly Inattentive Type; ADHD with Sleep Onset Insomnia; ADHD, ADD; ADHD, Predominantly Hyperactive - Impulsive; ADHD, Predominantly Inattentive Type; Hyperactivity; Hyperactivity Disorder; Inattention
Keywords: attention deficit hyperactivity disorder; attention deficit disorder; hyperactivity; inattention; adverse drug reaction; adverse events; side effects; nocebo effect; medication side effects; patient education; communication methods; communication strategies; pediatric care; parental satisfaction; pharmacological treatment; treatment; medication adherence; medication; child health; side effect management; treatment compliance; pediatric pharmacology; positive framing; negative framing; side effect reporting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Drug-Related Side Effects and Adverse Reactions; Medication Adherence; Patient Compliance

STUDY DESIGN:
Intervention Model Description: This study is a parallel-group randomized controlled care evaluation. This parallel design compares two already existing communication strategies regarding counseling on ADHD medication and adverse events in a clinical setting simultaneously. Random assignment to one of the two communication methods controls for potential biases and ensures that ob-served differences are attributable to the specific communication approach. A 4-week follow-up period is selected to provide adequate time for the medication's adverse events to become apparent and for meaningful data collection on adverse events and patient satisfaction.
  The study is planned to last a maximum period of 24 months. The anticipated start date is January 1st, 2025, with a projected end date no later than January 1st, 2027. Given that the pediatric department of the St. Antonius hospital sees more than 300 new ADHD patients an-nually and we aim to include 130 participants, we expect to complete the study within this timeframe.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Positively framed and concise information of adverse events (Experimental): PFI: A positively framed and concise discussion of adverse events (e.g. "Most children continue to feel fine with this medication, and if adverse events do occur, they often resolve quickly after the first few days of adjustment. If symptoms do appear, wait a little to see if they subside. If they persist and you are concerned, you can always check the package insert to see if it is listed as adverse event. You can also contact the clinic at any time."). A fixed script will be prepared for the treating paediatrician, and similar information will be provided in written form for parents and children.
  Interventions: Other: Communication Strategy for Side Effect Counseling in ADHD Treatment
- Negatively framed and comprehensive information of adverse events (Experimental): NFI: A comprehensive, negatively framed, discussion of the most common adverse events: difficulty falling asleep, decreased appetite, nausea, other gastrointestinal complaints, headache, sadness, or flat affect (e.g. "many patients experience nausea in the first month") as well as the more serious events like dullness of tics. A fixed script (see addendum) will be prepared for the treating paediatrician, and similar information will be provided to parents and their child in written form.
  Interventions: Other: Communication Strategy for Side Effect Counseling in ADHD Treatment

INTERVENTIONS:
Other: Communication Strategy for Side Effect Counseling in ADHD Treatment — One group receives negatively framed and extensive information about the most common adverse events of methylphenidate. A fixed script will be prepared for the treating paediatrician, and the same information will be provided in written form. The other group receives positively framed and concise information about the most common adverse events of methylphenidate. This information will also be provided in written form.

SUMMARY:
The goal of this randomized controlled care evaluation is to determine whether positively framed and concise information (PFI), compared to negatively framed and extensive information (NFI) about adverse events can reduce the number and severity of reported adverse events caused by ADHD medication in children aged 7 to 17 years. The main questions it aims to answer are:

1. Does PFI reduce the percentage of children suffering from decreased appetite in the first 4 weeks after starting medication compared to NFI?
2. Does PFI reduce the total number of adverse events compared to NFI?
3. Does PFI lower the total score on the Pittsburgh Side Effects Rating Scale (PSRS) compared to NFI?
4. Does PFI lead to higher parental satisfaction with the explanation of adverse events compared to NFI?
5. Does PFI reduce the number of patients who discontinue medication due to adverse events compared to NFI?
6. Does PFI decrease the number of patients needing melatonin for sleeping problems due to the use of methylphenidate compared to NFI?
7. What is the relationship between baseline factors such as age, ADHD or ADD diagnosis, and gender on the number of adverse events?

Researchers will compare children who receive positively framed, concise information (PFI) to those who receive negatively framed, detailed information (NFI) to determine if the framing of information affects the prevalence and severity of reported side effects, medication adherence, and parental satisfaction.

Participants in this study will:

* Be randomly assigned to receive either PFI or NFI about the side effects of methylphenidate.
* Start taking methylphenidate according to standard care protocols.
* Complete a Pittsburgh Side Effects Rating Scale (PSRS) questionnaire 4 weeks after starting medication to report any adverse events and their severity.
* Parents will provide feedback on satisfaction with the explanation of side effects using a short questionnaire.

This trial aims to inform best practices for communicating potential side effects to improve medication adherence and the overall treatment experience for children with ADHD and their families.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial designed to investigate the impact of positively framed information (PFI) versus negatively framed information (NFI) on the reporting of adverse events (AEs) associated with the initiation of methylphenidate treatment in children with ADHD or ADD. The trial aims to evaluate whether the manner in which information about side effects is communicated can influence the prevalence, severity, and perception of those side effects, as well as parental satisfaction and medication adherence.

Study Rationale Attention Deficit Hyperactivity Disorder (ADHD) is a highly prevalent childhood condition, with a global prevalence estimated between 5% and 5.5% (Polanczyk et al., 2014). This condition is defined by two main symptom categories: inattention and motor restlessness/impulsivity. These symptoms profoundly affect various aspects of a child's daily functioning (Carucci et al., 2020). Management of ADHD generally involves an integrated strategy that combines both pharmacological and non-pharmacological interventions (van der Schans et al., 2017).

Pharmacological treatment with stimulants such as methylphenidate and (lis-)dexamfetamine has been demonstrated to be highly effective, significantly reducing symptoms as reported by children and observed by parents and teachers (Cortese S et al., 2018 & Elliott et al., 2020). However, these treatments are often accompanied by adverse events (Elliott et al., 2020), with decreased appetite, abdominal pain, headaches and sleep disturbances being the most common, which can significantly impact the quality of life (Graham J et al., 2008 & Graham J et al., 2011). Adverse events of these medication most commonly lead to non-adherence to therapy, potentially resulting in long-term negative outcomes such as an increased risk of criminal behavior, substance abuse or traffic accidents (Kamimura-Nishimura et al., 2019). Evidence indicates that approximately 50% of children and adolescents fail to adhere to their prescribed treatment (Hodgkins et al., 2011). Therefore, minimizing adverse events to im-prove adherence to ADHD therapy is crucial.

According to the World Health Organization (2003), adherence is influenced by multiple fac-tors, including patient characteristics, the medical condition, therapy, the healthcare system, and socioeconomic circumstances. One factor that possibly influences the experience of ad-verse events in adults is the patient's expectation of experiencing them (Whitford et al., 2012 & Prediger et al., 2019 & Morris et al., 1982), which is partly shaped by the information provid-ed by healthcare professionals. These unintended expectation-induced adverse events are known as nocebo effects (Colloca et al., 2020). Studies in adults have shown that adverse events are more likely to occur if they are discussed beforehand, especially if presented neg-atively (e.g., "5% of the patients experience nausea") versus positively (e.g., "95% of the pa-tients do not experience nausea" or "95% feel well") (Webster et al., 2018 & Faase et al., 2019 & Smith et al., 2020). Moreover, studies have demonstrated that patients report more side effects following placebo treatment compared to those who are untreated (Colloca et al., 2020 & Howick et al., 2018 & Jensen et al., 2012 & Rief et al., 2011). Based on these and other studies, an expert group on placebo and nocebo mechanisms advised doctors to present information on treatments in such a way that nocebo effects are minimized (Evers et al 2021).

Despite extensive research on the nocebo effect in adults, studies specifically targeting chil-dren are virtually nonexistent. This is surprising given that children are naturally more sug-gestible than adults are and may possibly respond more strongly to both positively and nega-tively framed suggestions. Recent questionnaire-based research at our outpatient clinic, St. Antonius Hospital in the Netherlands (de Bruijn et al., 2023), indicated that parents and teen-agers prefer to receive positive information about potential adverse events. However, whether this indeed results in fewer adverse events in children is still unknown.

The primary objective of this study is to determine whether positively framed and concise in-formation (PFI), compared to negatively framed and extensive information (NFI) can reduce the number and severity of reported adverse events caused by ADHD medication in children aged 7 to 17 years. Secondary objectives are to assessing whether positively framed infor-mation can improve adherence to therapy by reducing the number or severity of adverse events and can reduce the need for melatonin due to sleeping problems. Previous research in adults has documented the impact of labeling and formulation on the occurrence of side ef-fects (Webster et al., 2018 & Faase et al., 2019 & Smith et al., 2020). However, similar studies in children are sparse. This study aims to bridge this gap by studying the extent to which ex-plicitly mentioning the potential for side effects influences their occurrence and severity in chil-dren, also known as the nocebo effect.

If positive language reduces the incidence or severity of side effects, this approach could be widely applied to a large group of patients in the Netherlands, potentially leading to better ad-herence to therapies and an improved quality of life. This might also reduce the necessity for additional medications like melatonin, which is commonly prescribed for sleep issues in this population, given that 25-50% of patients with attention-deficit hyperactivity disorder experi-ence sleep problems (Mohammadi et al., 2012). Moreover, positive outcomes from this study could prompt further research into the use of positive language with other commonly pre-scribed medications and patient groups, amplifying the overall impact. This study could also contribute to standardizing practices, as currently, there is a noticeable disparity among pedi-atricians treating ADHD patients-some provide extensive information about side effects, while others offer very little. Establishing a more uniform approach could enhance treatment consistency and outcomes.

Primary Objective To determine whether positively framed and concise information (PFI) reduces the percentage of children reporting decreased appetite in the first four weeks after starting methylphenidate compared to negatively framed and detailed information (NFI).

Secondary Objectives

1. To compare the total number and severity of reported adverse events between the PFI and NFI groups.
2. To assess the impact of PFI on parental satisfaction regarding the explanation of adverse events.
3. To evaluate whether PFI reduces the rate of medication discontinuation due to adverse events.
4. To determine whether PFI decreases the need for melatonin to manage sleep problems caused by methylphenidate.
5. To analyze the relationship between baseline factors (e.g., age, ADHD or ADD diagnosis, gender) and the number of reported adverse events.

Study Design This study is a parallel-group randomized controlled care evaluation. This parallel design compares two already existing communication strategies regarding counseling on ADHD medication and adverse events in a clinical setting simultaneously. Random assignment to one of the two communication methods controls for potential biases and ensures that ob-served differences are attributable to the specific communication approach. A 4-week follow-up period is selected to provide adequate time for the medication's adverse events to become apparent and for meaningful data collection on adverse events and patient satisfaction.

The study is planned to last a maximum period of 24 months. The anticipated start date is January 1st, 2025, with a projected end date no later than January 1st, 2027. Given that the pediatric department of the St. Antonius hospital sees more than 300 new ADHD patients annually and we aim to include 130 participants, we expect to complete the study within this timeframe. The primary workload involves reaching out to new patients and collecting follow-up questionnaires after 4 weeks.

Study Population Patients with ADHD or ADD, referred to the paediatric outpatient clinic of St. Antonius hospital, in the Utrecht region in the Netherlands and not yet using medication for AD(H)D will be invited to participate before their first consult with the paediatrician. This clinic serves a substantial number of new ADHD patients annually, providing a robust source population for the study. Given that the clinic sees over 300 new ADHD patients each year, recruiting 130 participants in 2 years seems highly feasible.

The study population will consist of children and adolescents aged 7 to 17 years, as this range encompasses the typical age for ADHD diagnosis and treatment. The study will aim for diversity in ethnic backgrounds, consistent with the clinic's patient base, to ensure that the findings are generalizable across different demographic groups. Participants will be newly diagnosed with ADHD and about to start medication.

Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Children aged 7 to 17 years
* Recently diagnosed with ADHD or ADD by a psychologist
* Desire to start ADHD/ADD medication expressed by both the child and the parents Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Previous use of stimulants
* 1st or 2nd degree family member using stimulants for ADHD/ADD within the last two years

Intervention

Prior to the consultation, randomization will occur between two communication methods:

1. NFI: A comprehensive, negatively framed, discussion of the most common adverse events: difficulty falling asleep, decreased appetite, nausea, other gastrointestinal complaints, headache, sadness, or flat affect (e.g. "many patients experience nausea in the first month") as well as the more serious events like dullness of tics. A fixed script (see addendum) will be prepared for the treating paediatrician, and similar information will be provided to parents and their child in written form.
2. PFI: A positively framed and concise discussion of adverse events (e.g. "Most children continue to feel fine with this medication, and if adverse events do occur, they often resolve quickly after the first few days of adjustment. If symptoms do appear, wait a little to see if they subside. If they persist and you are concerned, you can always check the package insert to see if it is listed as adverse event. You can also contact the clinic at any time."). A fixed script will be prepared for the treating paediatrician, and similar information will be provided in written form for parents and children.

Four weeks after starting the medication, a questionnaire will be sent out to systematically inquire about ADHD-related adverse events, assessing their occurrence and severity. Addi-tionally, parents and children will be asked to rate their satisfaction regarding the initial discus-sion about the condition, treatment explanation, and adverse event explanation using a 5-point Likert scale.

Outcome Measures The primary outcome measure is the percentage of children suffering from decreased appe-tite in the first 4 weeks of using methylphenidate. All adverse events and their severity will be assessed using the Pittsburgh Side-Effects Rating Scale (PSRS) (ref).

Secondary outcome measures are:

1. The total number of adverse events using the PSRS (0-14).
2. The total score on the PSRS (0-42)
3. Parental satisfaction with the communication on side effects with the physician on a scale from 0-4 (0= very unsatisfied, 1 = unsatisfied, 2 = neutral, 3 = satisfied, 4 = very satisfied).
4. The number of patients who have discontinued medication due to side effects.
5. the number of patients needing melatonine due to sleeping problems.

The association between factors such as age, ADHD or ADD diagnosis, gender, pre-existing sleeping problems, and medication dosage on the number of adverse events are considered as other study parameters.

Randomisation, blinding and treatment allocation Patients will be randomly allocated in a 1:1 ration to PFI or NFI after giving informed consent on the phone. They will be asked to bring the signed papers to the first consult. The treating pediatricians will be informed before the start of the consultation which script (PFI or NFI, see addendum) they have to use during the consult. The pediatricians are, therefore, not blinded. The results will be analyzed by a student who will be blinded for the randomisation. The ran-domisation will be perfomed by the research nurse (CB), who is not part of the study team.

Study procedures All children between 7 and 18 years, referred to the outpatient department of the St Antonius Hospital with a diagnosis of ADHD or ADD and a wish for starting ADHD~ medication will be invited to participate. The children will be seen by their paediatrician at baseline (either in the clinic or by a video consult, which is part of the standard care) and after 4-5 weeks after the start of the medication, to evaluate efficacy of the medication and discuss side effects. This is also standard care. The second consult can take place at the clinic, but also by phone. Just before visiting the paediatrician for the second time parents will be invited online to fill out, to-gether with their child, the PSRS as well as two short questions on satisfaction with the com-munication with the doctor and the pharmacy. The study ends after filling out these questions.

Safety Considerations This is a low-risk study involving two existing approaches to counseling on side effects. The burden on participants is minimal, as the interventions align with standard care practices. Participants retain the right to withdraw at any time, and adverse events will be managed according to standard clinical protocols.

Ethical Approval The study has been reviewed and approved by the Medical Ethics Committee-United (MEC-U) in the Netherlands. Informed consent is obtained from parents and, where applicable, children prior to participation.

Data Analysis All data will be analysed using SPSS under supervision of an epidemiologist. The dataset will be registered in an online data catalogue or web portal conform the FAIR principles. (Wil-kinson 2016). Data analysis will be performed according to the intention-to-treat principle. The intention to treat population will include all randomised patients, who will be analysed according to the group they are originally allocated to, despite of what treatment they have received. Furthermore, an additional analysis will be conducted in a per-protocol population.

Categorical variables will be expressed as a number with the percentage of the total alloca-tion arm. Continuous data with normal distribution will be reported as mean (standarddeviation) and continuous data without normal distribution as median (interquartile range).

Missing data will be addressed using appropriate statistical methods such as multiple imputa-tion or maximum likelihood estimation to ensure the integrity of the analysis. Participants with incomplete data on adverse events will be included in sensitivity analyses to assess the im-pact of missing data on the results.

Statistical analysis: a two-sided chi-square test with a significance level of 0.025 will be used for the statistical analysis of most of the outcome parameters. In addition, multiple regression analysis will be used to assess interaction effects of the different variables.

Potential Impact If positively framed information is shown to reduce the occurrence and severity of adverse events, this approach could standardize communication practices and improve medication adherence. The findings may also inform broader applications for other medications and patient populations.

Duration of Study Recruitment is expected to take approximately 10-12 months, with a total study duration of 24 months, including data analysis and dissemination of findings.

Dissemination Results will be published in peer-reviewed journals and presented at relevant national and international conferences. Findings will also be shared with clinical and academic organizations involved in ADHD care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 17 years
* Recently diagnosed with ADHD or ADD by a psychologist
* Desire to start ADHD/ADD medication expressed by both the child and the parents

Exclusion Criteria:

* Previous use of stimulants
* 1st or 2nd degree family member using stimulants for ADHD/ADD within the last two years

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events | From enrollment to 4 weeks after starting medication
  The primary outcome measure is the percentage of children suffering from decreased appetite in the first 4 weeks of using methylphenidate. All adverse events and their severity will be assessed using the Pittsburgh Side-Effects Rating Scale (PSRS).

SECONDARY OUTCOMES:
The total number of adverse events | From enrollment to 4 weeks after starting medication
  The total number of adverse events using the PSRS (0-14).
PSRS score | From enrollment to 4 weeks after starting medication
  The total score on the PSRS (0-42)
Parental satisfaction | From enrollment to 4 weeks after starting medication
  Parental satisfaction with the communication on side effects with the physician on a scale from 0-4 (0= very unsatisfied, 1 = unsatisfied, 2 = neutral, 3 = satisfied, 4 = very satisfied).
Patients who discontinued mediation | From enrollment to 4 weeks after starting medication
  The number of patients who have discontinued medication due to side effects.
Melatonine users | From enrollment to 4 weeks after starting medication
  The number of patients needing melatonine due to sleeping problems.

CONTACTS AND LOCATIONS:
Overall Officials: Arine Vlieger, MD, PhD, Principal Investigator — St. Antonius Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Waiting for central hub for databases for Dutch medical studies

REFERENCES:
- See also: 1. Colloca L, Barsky AJ. Placebo and nocebo effects. N Engl J Med [Internet]. 2020 [cited 2024 Sept 19];382(6):554-61. — http://dx.doi.org/10.1056/NEJMra1907805
- See also: 2. Kamimura-Nishimura KI, Brinkman WB, Froehlich TE. Strategies for improving ADHD medication adherence. Curr Psychiatry [Internet]. 2019 [cited 2024 Sept 19];18(8):25-38. — https://pubmed.ncbi.nlm.nih.gov/33867872/
- See also: Webster RK, Weinman J, Rubin GJ. Positively framed risk information in patient information leaflets reduces side effect reporting: A double-blind randomized controlled trial. Ann Behav Med [Internet]. 2018 [cited 2024 Sept 19];52(11):920-9. — https://pubmed.ncbi.nlm.nih.gov/30346496/
- See also: Polanczyk G, De Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry [Internet]. 2007 [cited 2024 Sept 20];164(6):942-8. Available from: https://pubmed.ncbi.nlm.ni — https://pubmed.ncbi.nlm.nih.gov/17541055/
- See also: Van Der Schans J, Çiçek R, Vardar S, Bos J, De Vries TW, Hoekstra PJ. Methylphenidate use and school performance among primary school children: a descriptive study. BMC Psychiatry [Internet]. 2017 [cited 2024 Sept 20];17. Available from: https://pubme — https://pubmed.ncbi.nlm.nih.gov/28356095/
- See also: Cortese S, Adamo N, Del Giovane C, Mohr-Jensen C, Hayes AJ, Carucci S, et al. Comparative efficacy and tolerability of medications for attention-deficit hyperactivity disorder in children, adolescents, and adults: a systematic review and network meta — http://dx.doi.org/10.1016/S2215-0366(18)30269-4
- See also: Elliott J, Johnston A, Husereau D, Kelly SE, Eagles C, Charach A, et al. Pharmacologic treatment of attention deficit hyperactivity disorder in adults: A systematic review and network meta-analysis. PLoS One [Internet]. 2020 [cited 2024 Sept 20];15(1 — http://dx.doi.org/10.1371/journal.pone.0240584
- See also: NICE. Attention deficit hyperactivity disorder (update). [C] Evidence reviews for pharmacological efficacy and sequencing pharmacological treatment. NICE guideline [Internet]. September 2017 [cited 2024 Sep 20]; Available from: https://www.nice.org.u — https://www.nice.org.uk/guidance/indevelopment/gid-cgwave0798
- See also: Nanda A, Janga LSN, Sambe HG, Yasir M, Man RK, Gogikar A, et al. Adverse effects of stimulant interventions for attention deficit hyperactivity disorder (ADHD): A comprehensive systematic review. Cureus [Internet]. 2023 [cited 2024 Sept 20];15(9):e45 — http://dx.doi.org/10.7759/cureus.45995
- See also: Kamal M, Eltohami M, Al-Shibli S. Effect and side effect of stimulant/methylphenidate on children and adolescents with ADHD: the Qatar experience. Arch Pediatr [Internet]. 2018 [cited 2024 Sept 20];3:160. Available from: https://www.gavinpublishers.c — https://www.gavinpublishers.com/article/view/effect-and-side-effect-of-stimulant-methylphenidate-on-children-and-adolescents-with-adhd-the-qatar-experience
- See also: Graham J, Coghill D. Adverse effects of pharmacotherapies for attention-deficit hyperactivity disorder: epidemiology, prevention and management. CNS Drugs [Internet]. 2008 [cited 2024 Sept 20];22(3):213-37. Available from: https://pubmed.ncbi.nlm.nih — https://pubmed.ncbi.nlm.nih.gov/18278977/
- See also: Hodgkins P, Sasané R, Christensen L, Harley C, Liu F. Treatment outcomes with methylphenidate formulations among patients with ADHD: retrospective claims analy-sis of a managed care population. Curr Med Res Opin [Internet]. 2011 [cited 2024 Sept 20]; — https://pubmed.ncbi.nlm.nih.gov/21973231/
- See also: World Health Organization. Adherence to long-term therapies: Evidence for action. Genève, Switzerland: World Health Organization [Internet]. 2003 [cited 2024 Sept 20]. Available from: https://iris.who.int/handle/10665/42682 — https://iris.who.int/handle/10665/42682
- See also: Whitford HS, Olver IN. When expectations predict experience: the influence of psychological factors on chemotherapy toxicities J. J Pain Symptom Manage [Internet]. 2012 [cited 2024 Sept 23];43(6):1036-50. Available from: https://pubmed.ncbi.nlm.nih.g — https://pubmed.ncbi.nlm.nih.gov/22651947/
- See also: Prediger B, Meyer E, Büchter R, Mathes T. Nocebo effects of a simplified package leaflet compared to unstandardised oral information and a standard package leaflet: a pilot randomised controlled trial. Trials [Internet]. 2019 [cited 2024 Sept 23];20( — http://dx.doi.org/10.1186/s13063-019-3565-3
- See also: De Bruijn C, Hamming G, Knibbe C, Tromp E, Benninga MA. Vlieger AM. Teenagers' and parental individual needs for side effects information and the influence of nocebo effect education. Patient Educ Couns [Internet]. 2023 [cited 2024 Sept 23];108(10758 — https://pubmed.ncbi.nlm.nih.gov/36516654/
- See also: Mohammadi MR, Mostafavi SA, Keshavarz SA, Eshraghian MR, Hosseinzadeh P, Hosseinzadeh-Attar MJ, et al. Melatonin effects in methylphenidate treated children with attention deficit hyperactivity disorder: a randomized double blind clinical trial. Iran — https://pubmed.ncbi.nlm.nih.gov/22952551/
- See also: Lee J, Grizenko N, Bhat V, Sengupta S, Polotskaia A, Joober R. Relation between therapeutic response and side effects induced by methylphenidate as observed by parents and teachers of children with ADHD. BMC Psychiatry [Internet]. 2011 [cited 2024 Se — http://dx.doi.org/10.1186/1471-244X-11-70
- See also: Wilkinson M, Dumontier M, Aalbersberg I. The FAIR guiding principles for scien-tific data management and stewardship. Sci Data [Internet]. 2016 [cited 2024 Sept 25]; 3. Available from: https://pubmed.ncbi.nlm.nih.gov/26978244/ — https://pubmed.ncbi.nlm.nih.gov/26978244/